CLINICAL TRIAL: NCT02650518
Title: Controlling Antimicrobial Use Through Reducing Unnecessary Treatment of Catheter Associated Urinary Tract Infections (CARCUTI)
Brief Title: Controlling Antimicrobial Use Through Reducing Unnecessary Treatment of Catheter Associated Urinary Tract Infections
Acronym: CARCUTI
Status: Unknown | Phase: Phase 2 / Phase 3 | Type: Interventional
Last Known Status: Recruiting
Sponsor: National University Hospital, Singapore (Other)
Collaborators: Tan Tock Seng Hospital (Other); Singapore General Hospital (Other); National University of Singapore (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 2014/00589
Record Dates: First submitted 2015-12-30; First posted 2016-01-08 (Estimated); Last update posted 2016-01-08 (Estimated); Status verified 2016-01

CONDITIONS: Catheter-Related Infections
Keywords: Catheter-Associated Urinary Tract Infections; Antimicrobial Stewardship; Short-Course Antimicrobials
MeSH Terms: conditions — Catheter-Related Infections

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Control (No Intervention): Subject receives the standard of care that is provided by the primary team taking up his/her case.
- Catheter change+Short-course Antibiotics (Experimental)
  Interventions: Other: Short-course Antibiotics; Device: Catheter Change

INTERVENTIONS:
Other: Short-course Antibiotics — 3 days of amoxicillin/clavulanate, ciprofloxacin, or cotrimoxazole.
  Arms: Catheter change+Short-course Antibiotics
Device: Catheter Change — Urinary catheter change once randomization is complete.
  Arms: Catheter change+Short-course Antibiotics

SUMMARY:
Hypothesis: A short course (3-5 days) of antibiotic therapy (experimental arm) is as safe and effective as a long course of antibiotic therapy for the treatment of catheter-associated urinary tract infections.

ELIGIBILITY:
Inclusion Criteria:

1. Inpatients ≥ 21 years old.
2. Presence of indwelling urinary catheter at the time of urine culture for ≥2days.
3. Fever >38°C.
4. A urine specimen sent to the hospital microbiological laboratory for culture.
5. An antibiotic order for presumed symptomatic catheter associated urinary tract infection.

Exclusion Criteria:

1. Persistent fever >38°C for more than 24 hours, or any fever >38.9°C.
2. Haemodynamic instability, defined as:

   * Requirement for intravenous vasopressor agents
   * Systolic blood pressure <90 mmHg
   * Acute hypotensive event with drop in systolic blood pressure of >30 mmHg or diastolic blood pressure of >20 mmHg
3. The following laboratory values within the previous 48 hours (if available):

   * White blood cell count>15 or <4 x10^9/L.
   * Procalcitonin>0.25ug/mL
   * C Reactive Protein >100mg/mL
   * An increase in the serum creatinine of more than 50% from baseline
4. New requirement for oxygen supplement.
5. Current admission to a high dependency unit or ICU.
6. Radiological evidence of an upper urinary tract infection
7. Flank pain or tenderness, suggesting an upper urinary tract infection
8. Urologic surgical procedure within the previous 72 hours
9. Known structural genitourinary abnormalities including:

   * Nephrostomy tubes
   * Tumours of the urinary tract
   * Ureteric stenting
   * Ureteric strictures
   * Urolithiasis
10. Bloodstream or other significant infection suspected at any site other than the catheterized urinary tract.
11. Received antibiotics for more than 48 hours prior to randomization.
12. Positive urinary culture with organism resistant to all the investigational antibiotics in the week prior to randomisation.
13. Hypersensitivity to ciprofloxacin, cotrimoxazole and amoxicillin-clavulanate.
14. Pregnancy.

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 500 (Estimated)
Dates: Start 2015-12; Primary Completion 2017-10 (Estimated); Study Completion 2018-10 (Estimated)

PRIMARY OUTCOMES:
Resolution | Day 14 post-randomisation
  Resolution of signs and symptoms of CAUTI

SECONDARY OUTCOMES:
Short-Term Resolution | day 3 and day 7 post-randomisation
  Resolution of signs and symptoms of CAUTI
Recurrence of fever or symptoms | 7, 14 and 30 days post randomization
Haemodynamic instability | day 14 post randomization
Admission to high dependency or intensive care units | 14 days post-randomization
Length of hospitalization | 30 days post-randomization
Re-admission | Day 30 post-randomization
Secondary Infections | 3 months post-randomization
Recurrent Urinary Tract Infections | 3 months and 1 year post-randomization
Urologic surgery or procedure | 1 year post-randomization
Antimicrobial use and duration | 1 month post-randomization
Colonization or infection by antibiotic-resistant organisms | 30 days post-randomization

CONTACTS AND LOCATIONS:
Overall Officials: Paul A Tambyah, MD, Principal Investigator — National University Hospital, Singapore
Locations (3):
- Singapore (3):
  - National University Hospital, Singapore
  - Singapore General Hospital, Singapore
  - Tan Tock Seng Hospital, Singapore

REFERENCES:
- [Background] Edwards JR, Peterson KD, Andrus ML, Tolson JS, Goulding JS, Dudeck MA, Mincey RB, Pollock DA, Horan TC; NHSN Facilities. National Healthcare Safety Network (NHSN) Report, data summary for 2006, issued June 2007. Am J Infect Control. 2007 Jun;35(5):290-301. doi: 10.1016/j.ajic.2007.04.001. No abstract available. PMID 17577475
- [Background] Schaberg DR, Weinstein RA, Stamm WE. Epidemics of nosocomial urinary tract infection caused by multiply resistant gram-negative bacilli: epidemiology and control. J Infect Dis. 1976 Mar;133(3):363-6. doi: 10.1093/infdis/133.3.363. No abstract available. PMID 768384
- [Background] Milan PB, Ivan IM. Catheter-associated and nosocomial urinary tract infections: antibiotic resistance and influence on commonly used antimicrobial therapy. Int Urol Nephrol. 2009;41(3):461-4. doi: 10.1007/s11255-008-9468-y. Epub 2008 Sep 12. PMID 18787972
- [Background] Tambyah PA, Knasinski V, Maki DG. The direct costs of nosocomial catheter-associated urinary tract infection in the era of managed care. Infect Control Hosp Epidemiol. 2002 Jan;23(1):27-31. doi: 10.1086/501964. PMID 11868889
- [Background] Wald HL, Ma A, Bratzler DW, Kramer AM. Indwelling urinary catheter use in the postoperative period: analysis of the national surgical infection prevention project data. Arch Surg. 2008 Jun;143(6):551-7. doi: 10.1001/archsurg.143.6.551. PMID 18559747
- [Background] Hooton TM, Bradley SF, Cardenas DD, Colgan R, Geerlings SE, Rice JC, Saint S, Schaeffer AJ, Tambayh PA, Tenke P, Nicolle LE; Infectious Diseases Society of America. Diagnosis, prevention, and treatment of catheter-associated urinary tract infection in adults: 2009 International Clinical Practice Guidelines from the Infectious Diseases Society of America. Clin Infect Dis. 2010 Mar 1;50(5):625-63. doi: 10.1086/650482. PMID 20175247
- [Background] Ng E, Earnest A, Lye DC, Ling ML, Ding Y, Hsu LY. The excess financial burden of multidrug resistance in severe gram-negative infections in Singaporean hospitals. Ann Acad Med Singap. 2012 May;41(5):189-93. PMID 22760715
- [Background] Harding GK, Nicolle LE, Ronald AR, Preiksaitis JK, Forward KR, Low DE, Cheang M. How long should catheter-acquired urinary tract infection in women be treated? A randomized controlled study. Ann Intern Med. 1991 May 1;114(9):713-9. doi: 10.7326/0003-4819-114-9-713. PMID 2012351
- [Background] Peterson J, Kaul S, Khashab M, Fisher AC, Kahn JB. A double-blind, randomized comparison of levofloxacin 750 mg once-daily for five days with ciprofloxacin 400/500 mg twice-daily for 10 days for the treatment of complicated urinary tract infections and acute pyelonephritis. Urology. 2008 Jan;71(1):17-22. doi: 10.1016/j.urology.2007.09.002. PMID 18242357
- [Background] Dow G, Rao P, Harding G, Brunka J, Kennedy J, Alfa M, Nicolle LE. A prospective, randomized trial of 3 or 14 days of ciprofloxacin treatment for acute urinary tract infection in patients with spinal cord injury. Clin Infect Dis. 2004 Sep 1;39(5):658-64. doi: 10.1086/423000. Epub 2004 Aug 13. PMID 15356779
- [Background] Raz R, Schiller D, Nicolle LE. Chronic indwelling catheter replacement before antimicrobial therapy for symptomatic urinary tract infection. J Urol. 2000 Oct;164(4):1254-8. PMID 10992375
- [Background] Darouiche RO, Al Mohajer M, Siddiq DM, Minard CG. Short versus long course of antibiotics for catheter-associated urinary tract infections in patients with spinal cord injury: a randomized controlled noninferiority trial. Arch Phys Med Rehabil. 2014 Feb;95(2):290-6. doi: 10.1016/j.apmr.2013.09.003. Epub 2013 Sep 11. PMID 24035770
- [Background] Singh N, Rogers P, Atwood CW, Wagener MM, Yu VL. Short-course empiric antibiotic therapy for patients with pulmonary infiltrates in the intensive care unit. A proposed solution for indiscriminate antibiotic prescription. Am J Respir Crit Care Med. 2000 Aug;162(2 Pt 1):505-11. doi: 10.1164/ajrccm.162.2.9909095. PMID 10934078
- [Background] Hamasuna R, Takahashi S, Yamamoto S, Arakawa S, Yanaihara H, Ishikawa S, Matsumoto T. Guideline for the prevention of health care-associated infection in urological practice in Japan. Int J Urol. 2011 Jul;18(7):495-502. doi: 10.1111/j.1442-2042.2011.02769.x. Epub 2011 May 16. PMID 21569109
- [Background] Tambyah PA, Maki DG. Catheter-associated urinary tract infection is rarely symptomatic: a prospective study of 1,497 catheterized patients. Arch Intern Med. 2000 Mar 13;160(5):678-82. doi: 10.1001/archinte.160.5.678. PMID 10724054
- [Background] Corey GR, Stryjewski ME. New rules for clinical trials of patients with acute bacterial skin and skin-structure infections: do not let the perfect be the enemy of the good. Clin Infect Dis. 2011 Jun;52 Suppl 7:S469-76. doi: 10.1093/cid/cir162. PMID 21546623
- [Background] Blackwelder WC. "Proving the null hypothesis" in clinical trials. Control Clin Trials. 1982 Dec;3(4):345-53. doi: 10.1016/0197-2456(82)90024-1. PMID 7160191
- [Background] Scott IA. Non-inferiority trials: determining whether alternative treatments are good enough. Med J Aust. 2009 Mar 16;190(6):326-30. doi: 10.5694/j.1326-5377.2009.tb02425.x. PMID 19296815